CLINICAL TRIAL: NCT03342248
Title: Evaluation of the Impact of a Social Network Via a Digital Platform for Caregivers of Patients Suffering From Mental Disorders
Acronym: CONNECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-17
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- access to the social network (Experimental): This group is made up of carers who have access to the social network via a digital platform developed during step 1. This network will offer features from step 1 (sharing experiences on a forum, monitoring health status )
  Interventions: Other: access to the social network
- no access to the network (No Intervention): This group consists of caregivers who do not have access to the social network via a digital platform developed during step 1.
  Access to the social network will be offered to all carers at the end of the study, especially those assigned in the control group to limit their refusal to participate.

INTERVENTIONS:
Other: access to the social network — The development of a social network via a digital platform for carers of patients suffering from severe mental illness and study of the impact of its use on the health status of caregivers
  Arms: access to the social network

SUMMARY:
Severe mental illnesses have a significant social cost, as much by their impact on the sick as on their entourage. The Deinstitutionalization and care in the community of patients with severe mental illness result in increased families and loved ones (also known as "informal caregivers" or "informal caregivers") If psychoeducation programs have been developed to help caregivers better manage and cope with the illness of the person being helped (optimize the quality of care, manage anxiety and isolation, these initiatives appear minimal in view of the magnitude of the burden (notion of burden: "burden") and the suffering of caregivers. Quality of life levels remain extremely low compared to the general population, nearly 4 out of 10 caregivers show a sense of inability to cope with the "permanent anxiety" of this load, 1/3 feels depressed and over 1/10 feels isolated on a personal and professional level

DETAILED DESCRIPTION:
This project will take place in three stages:

1- Development and development of the network: the conception of the social network is based on the point of view of the caregivers, which is one of the originalities of this project. Current social networks are very "medico-centric" And often poorly adapted to the needs of caregivers of patients suffering from pathologies mental disorders. This step is based on a qualitative approach to these caregivers. Focus groups (5 focus of 5 carers) will be led by a psychologist in order to understand their experience and identify the resulting needs in order to determine the architecture and services offered on the network social. From emerging needs, a study based on Delphi method will be conducted with professionals from different disciplines psychiatry, public health, communication and information professionals, ethicists, health economists and sociologists) to provide a light on the professional responses that can be proposed to the needs of carers. The development of the social network will be done in close collaboration with a caregiver who will be in charge of the animation and moderation of the network 2. Implementation of the randomized trial comparing two groups of caregivers (access to the social network vs. lack of access to the social network) over a period of 6 month. The same scales will be filled by both groups at T0 and then at 6 months.

3. Qualitative approach to network perception: semidirective interviews made by a psychologist to a panel of caregivers using the network at course of 6 months

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of patient suffering from a severe mental illness and consultant in one of the investigative centers
* over 18 years old
* Caregiver who has no problem understanding current French Careguiver who has agreed to participate in the study. The definition of the caregiver is that given by the High Authority of Health (HAS): The so-called natural caregivers are the unprofessional people who come to the help of a person dependent on his entourage for the activities of daily life.

Exclusion Criteria:

* Minors caregivers
* not speaking and not reading enough French to participate in the study
* not having agreed to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2018-02-02 (Estimated); Primary Completion 2020-02-02 (Estimated); Study Completion 2020-09-02 (Estimated)

PRIMARY OUTCOMES:
quality of life | Baseline
  The quality of life of caregivers is assessed using a specific questionnaire , validated, designed to measure the quality of life of caregivers.
  caregivers of patients suffering from mental pathology: the CGSQoL (Auquier 2013). This questionnaire has satisfactory psychometric properties and is sensitive to change.

SECONDARY OUTCOMES:
Quality of life | 6 months
  The quality of life of caregivers is assessed using a specific questionnaire , validated, designed to measure the quality of life of caregivers.
  caregivers of patients suffering from mental pathology: the CGSQoL (Auquier 2013). This questionnaire has satisfactory psychometric properties and is sensitive to change.
self-administered questionnaires | 6 months
  Zarit's scale

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Conception, Marseille, France